CLINICAL TRIAL: NCT00698035
Title: A Phase II Study of Vaginal Testosterone Cream vs. the ESTRING for Vaginal Dryness or Decreased Libido in Early Breast Cancer Patients Treated With Aromatase Inhibitors
Brief Title: Vaginal Testosterone Cream vs ESTRING for Vaginal Dryness or Decreased Libido in Early Stage Breast Cancer Patients
Acronym: E-String
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCSF-067519
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Sexual Dysfunction, Physiological
Keywords: Vaginal Testosterone Cream; ESTRING
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone Cream (Active Comparator): Testosterone Cream 1% micronized in velvachol - 0.5 gm of cream vaginally each night for two weeks, then 3 times a week for total of 12 weeks of treatment
  Interventions: Drug: Testosterone Cream
- Estring (Active Comparator): Estring 2mg ring inserted vaginally once every 12 weeks
  Interventions: Drug: Estring

INTERVENTIONS:
Drug: Testosterone Cream — 1% micronized in velvachol - 0.5 gm of cream vaginally each night for two weeks, then 3 times a week for total of 12 weeks of treatment
  Other Names: intravaginal testosterone cream
  Arms: Testosterone Cream
Drug: Estring — 2mg ring inserted vaginally once every 12 weeks
  Other Names: ESTRING Estrodial Vaginal Ring
  Arms: Estring

SUMMARY:
The purpose of this clinical research study is to determine whether the ESTRING or a special preparation of a testosterone cream inserted vaginally are safe for use in breast cancer patients. This study will also evaluate if either of these treatments can improve symptoms of vaginal dryness or decreased sexual interest that are related to your treatment for breast cancer.

DETAILED DESCRIPTION:
There is a growing body of scientific literature to suggest that sexual functioning is one of the most distressing problems experienced by breast cancer survivors. Vaginal dryness, dyspareunia (pain during sexual intercourse), and decreased libido are common complaints among breast cancer patients. With increasing use of aromatase inhibitors which are associated with a higher rate of vaginal dryness than tamoxifen, these problems are becoming even more prominent. This study will evaluate the safety and tolerability of the ESTRING and 1% testosterone cream administered vaginally as treatments for vaginal dryness and/or decreased libido in women receiving an aromatase inhibitor for early stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed Stage I-III breast cancer who are taking an aromatase inhibitor as adjuvant hormonal therapy. Patient must have started the aromatase inhibitor at least 60 days prior to enrolling.
2. Postmenopausal estradiol levels at baseline as measured by standard laboratory analysis.

   * Patient may be rendered postmenopausal through the use of a GnRH agonist, but must have confirmed post-menopausal levels of serum estradiol on two lab tests at least one month apart.
   * If patient has been rendered post-menopausal by adjuvant chemotherapy but has had a period within the past 12 months, post-menopausal levels of serum estradiol must be documented on two lab tests at least 3 months apart.
3. Age ≥18 and ≤80 years old.
4. ECOG ≤1
5. Adequate hematologic, hepatic, and renal function as defined by:

   * Hgb ≥9 g/dL
   * Absolute neutrophil count (ANC)/absolute granulocyte count (AGC) ≥1500 cells/mm3
   * Platelet count ≥100,000/mm3
   * Serum creatinine ≤1.5 mg/dL
   * Total bilirubin ≤1.5 times the ULN; and aspartate aminotransferase ≤3 times the ULN
6. Normal thyroid function tested within the past 6 months (Patients with a diagnosis of hypothyroidism and on thyroid supplementation must have had thyroid function tests in the normal range within the past 3 months)
7. Patient must have recovered from the side effects of previous chemotherapy, surgery, or radiation therapy for early breast cancer.

Exclusion Criteria:

1. History of radiation to the vaginal area
2. Concurrent treatment with any type of oral, injectable or topical form of estrogen or androgen therapy including natural supplements marketed as hormone replacement products
3. Initiation of topical moisturizers (for example, Replens), or herbal or alternative medicines to manage the symptoms of vaginal dryness while on study. Patients who were previously using these products may continue them with the same usage pattern while on study.
4. Use of vaginal hormonal products (rings, inserts, creams, gels) containing estrogens or androgens within the past 30 days.
5. History of an abnormal pap smear within the last 12 months
6. History of endometrial or ovarian cancer
7. Any episode of vaginal bleeding in the past 6 months that has not been evaluated by a gynecological exam and/or pelvic ultrasound
8. History of sexual dysfunction prior to diagnosis of breast cancer ( Sexual dysfunction will be defined as loss of libido or inability to achieve orgasm for which patient sought medical attention or which patient felt significantly interfered with quality of life.)
9. Moderate or severe depression for which the patient is receiving ongoing psychological counseling and/or taking antidepressants, and for whom, in the investigators opinion may be interfering in the patients sexual function independent of the side effects of breast cancer and aromatase inhibitor use.
10. Use of any investigational agent for breast cancer within 3 weeks of study entry.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-03; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Melisko, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Derived] Melisko ME, Goldman ME, Hwang J, De Luca A, Fang S, Esserman LJ, Chien AJ, Park JW, Rugo HS. Vaginal Testosterone Cream vs Estradiol Vaginal Ring for Vaginal Dryness or Decreased Libido in Women Receiving Aromatase Inhibitors for Early-Stage Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2017 Mar 1;3(3):313-319. doi: 10.1001/jamaoncol.2016.3904. PMID 27832260

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 76 enrolled participants, one participant consented and was assigned to ESTRING, but did not insert ESTRING prior to withdrawing from the study.
Period: Overall Study
Arm/Group | Estring | Testosterone Cream
Started | 39 | 36
Completed | 35 | 34
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics for 75 participants who initiated treatment. One participant consented and was assigned to ESTRING, but did not insert ESTRING prior to withdrawing from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Estring | Testosterone Cream | Total
Number analyzed (Participants) | 39 | 36 | 75
Age, Continuous [Mean (Full Range); unit: years] | 56 [37 to 78] | 57 [38 to 74] | 56 [37 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 75
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 36 | 75

OUTCOME MEASURES:

1. Secondary Outcome: Serum Estradiol (E2)
Description: serial measurements of serum estradiol (E2) by liquid chromatography tandem mass spectrometry (Quest Diagnostics)
Time Frame: 12 weeks
Population: Per protocol, participants who completed 12 weeks of assigned treatment
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Estring | Testosterone Cream
Number analyzed (Participants) | 35 | 34
pg/ml
  E2 at baseline | 27 (36) | 9 (13)
  E2 at 4 weeks | 5 (5) | 10 (20)
  E2 at 12 weeks | 9 (12) | 8 (7)

2. Secondary Outcome: Matched E2 by Commercial and Research (RIA) Analyses
Description: Serum estradiol assays sent to the UCSF clinical laboratory are sent out to Quest Diagnostics, which uses LC/MS for their ultra-sensitive estradiol assay. Samples were also sent to a specialized research lab in England which has developed an ultrasensitive assay using radioimmunoassay (RIA) after ether extraction (sensitivity limit of 3pmol/l) to quantify low levels of estradiol found in post-menopausal women
Time Frame: baseline, 4 weeks
Population: Patients from both study arms arms with matched pairs of baseline and week 4 E2 performed by both commercial and research labs
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- E2 by LC/MS: A commercially available ultrasensitive E2 level was measured at baseline and 4 weeks (Quest Diagnostics, liquid chromatography tandem mass spectrometry (LC/MS, PM range <10 pg/ml)
- E2 by RIA: Additional measurement of baseline and week 4 E2 by RIA
Arm/Group | E2 by LC/MS | E2 by RIA
Number analyzed (Participants) | 63 | 63
pg/ml
  Baseline E2 | 17.7 (28.5) | 17.9 (44.1)
  4-week E2 | 7.8 (15.0) | 2.9 (13.4)
Statistical Analysis 1: Comparison: E2 by LC/MS vs E2 by RIA; Comparison of baseline estradiol between LC/MS and RIA; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Significant at p<0.05
Statistical Analysis 2: Comparison: E2 by LC/MS vs E2 by RIA; Comparison of week 4 estradiol between LC/MS and RIA; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — singificant at p<0.05

3. Primary Outcome: Persistently Elevated Serum Estradiol Level Outside the Post-menopausal Range
Description: Liquid chromatography tandem mass spectrometry (Quest Diagnostics). Persistently elevated serum estradiol level outside the post-menopausal range was defined as: Serum estradiol >10 pg/dl on two consecutive collections at least 4 weeks apart. 2. If baseline estradiol was >10 pg/dl, subsequent levels >10 pg/ml higher than baseline were considered a significant elevation outside the post-menopausal range.
Time Frame: 12 Weeks
Population: Per protocol, to be considered evaluable for the Primary Outcome, patients must complete both baseline evaluation and week 4 safety blood draw. 1 participant in the Testosterone arm was not evaluable.
Measure: Number; unit: participants
Arm/Group | Estring | Testosterone Cream
Number analyzed (Participants) | 35 | 33
participants | 0 | 4

4. Secondary Outcome: Total Testosterone Levels
Description: By serum ultrasensitive total testosterone test (Quest Diagnostics)
Time Frame: 12 weeks
Population: Per protocol, participants assigned to the Testosterone arm who completed 12 weeks of assigned treatment and had testosterone measurement at baseline, 4 weeks and 12 weeks.
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Testosterone Cream
Number analyzed (Participants) | 27
ng/dl
  Testosterone at baseline | 33 (19)
  Testosterone at 4 weeks | 186 (276)
  Testosterone at 12 weeks | 171 (251)

5. Secondary Outcome: Sexual Quality of Life
Description: Cancer Rehabilitation Evaluation System (CARES) Sexual Dysfunction (SD) and Sexual Interest (SI) Subscales range from 0 to 4 and measure the severity of problems, with higher scores indicating more difficulty.
Time Frame: Baseline, Week 4, Week 12
Population: Participants who provided responses to SD, SI and SS at 3 time points: Baseline (BL), Week 4 (W4), and Week 12 (W12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Estring | Testosterone Cream
Number analyzed (Participants) | 32 | 30
units on a scale
  SI (BL) | 1.2 (0.9) | 1.4 (0.8)
  SI (W4) | 1.3 (1.0) | 1.2 (0.7)
  SI (W12) | 0.9 (0.7) | 1.0 (0.6)
  SD (BL) | 2.9 (1.1) | 2.9 (0.8)
  SD (W4) | 2.4 (1.1) | 2.1 (1.0)
  SD (W12) | 2.0 (1.1) | 1.9 (1.1)
Statistical Analysis 1: Comparison: Estring; Change in SI from BL to W12; Test type: Superiority or Other; p = 0.021, t-test, 2 sided — Significant at p<0.05
Statistical Analysis 2: Comparison: Estring; Change in SD from BL to W12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Significant at p<0.05
Statistical Analysis 3: Comparison: Testosterone Cream; Change in SI from BL to W12; Test type: Superiority or Other; p = 0.0228, t-test, 2 sided — Significant at p<0.05
Statistical Analysis 4: Comparison: Testosterone Cream; Change in SD from BL to W12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Significant at p<0.05

6. Secondary Outcome: Sexual Satisfaction
Description: Participants were asked to respond to a Sexual Satisfaction One Item Measure which asked "Overall, how satisfactory to you is your sexual relationship with your partner?" Response options range from 1 (Extremely unsatisfactory) to 6 (Extremely satisfactory).
Time Frame: Baseline, Week 4, Week 12
Population: Participants who provided responses to SD, SI and SS at all 3 time points: Baseline (BL), Week 4 (W4), and Week 12 (W12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Estring | Testosterone Cream
Number analyzed (Participants) | 32 | 30
units on a scale
  SS (BL) | 2.5 (1.6) | 3.2 (1.6)
  SS (W4) | 3.5 (1.8) | 3.7 (1.6)
  SS (W12) | 4.0 (1.5) | 4.0 (1.5)
Statistical Analysis 1: Comparison: Estring; Change in SS from Baseline to Week 12; Test type: Superiority or Other; p = 0.004, t-test, 2 sided — Significant at p<0.05
Statistical Analysis 2: Comparison: Testosterone Cream; Change in SS from Baseline to Week 12; Test type: Superiority or Other; p = 0.139, t-test, 2 sided — Significant at p<0.05

7. Secondary Outcome: Change in Vaginal Epithelium Scores
Description: During a gynecologic exam, the vaginal epithelium was assessed by an examiner using the Vaginal Atrophy Scoring Scale to evaluate Rugae (lack of), Pallor (pinkness), Petechiae, Mucosal thinning, Dryness. Scores range from 0 (none) to 3 (severe); higher scores indicate less favorable outcomes.
Time Frame: Baseline, 12 weeks
Population: Patients with both baseline and week 12 gynecologic exams for evaluation of vaginal atrophy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Estring | Testosterone Cream
Number analyzed (Participants) | 35 | 34
units on a scale
  Rugae | -1.03 (0.80) | -0.71 (0.84)
  Pallor | -0.88 (0.84) | -0.91 (0.75)
  Petechiae | -1.0 (1.07) | -0.74 (1.38)
  Mucosal thinning | -0.62 (0.49) | -0.88 (0.64)
  Dryness | -1.03 (0.80) | -0.71 (0.91)
Statistical Analysis 1: Comparison: Estring; Differences in rugae, pallor, petechiae, mucosal thinning and dryness between baseline and week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Significant at p<0.05
Statistical Analysis 2: Comparison: Testosterone Cream; Differences in rugae, pallor, mucosal thinning, and dryness from baseline to 12 weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Significant at p<0.05
Statistical Analysis 3: Comparison: Testosterone Cream; Difference in petechiae between baseline and week 12; Test type: Superiority or Other; p = 0.0061, t-test, 2 sided — Significant at p<0.05

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Estring | Testosterone Cream
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/36
Other Adverse Events (participants affected / at risk) | 10/39 | 10/36
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estring (N=39) | Testosterone Cream (N=36)
Vaginal discharge (Reproductive system and breast disorders) | 4 (4) | 2 (2)
Facial hair growth (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Hot flashes (General disorders) | 3 (3) | 1 (1)
Vaginal itching or irritation (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Vaginal odor (Reproductive system and breast disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes